CLINICAL TRIAL: NCT03590652
Title: Phase II Study of the Combination of Daratumumab, Ixazomib, Pomalidomide, and Dexamethasone as Salvage Therapy in Relapsed/Refractory Multiple Myeloma A University of California Hematologic Malignancies Consortium Protocol (UCHMC1809)
Brief Title: Daratumumab, Ixazomib, Pomalidomide, and Dexamethasone as Salvage Therapy in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial met its primary endpoint.
Sponsor: University of California, San Diego (Other)
Collaborators: Celgene (Industry); Takeda (Industry); Janssen, LP (Industry)
Responsible Party: Principal Investigator, Caitlin Costello, MD, Associate Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180638
Record Dates: First submitted 2018-06-21; First posted 2018-07-18 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: multiple myeloma; relapsed/refractory multiple myeloma; Daratumumab; Pomalidomide; Ixazomib; Dexamethasone; cancer; Phase 2; Darzalex; Pomalyst; Ninlaro; Decadron
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — ixazomib; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ixazomib, daratumumab, pomalidomide and dexamethasone (Experimental): Daratumumab will be administered at 16mg/kg IV weekly x 8 weeks, biweekly x 8 weeks, then monthly. Pomalidomide 4mg will be administered orally daily for days 1-21. Patients ≤ age 75 will receive a 40mg dose of dexamethasone, and those over the age of 75 may receive a 20mg dose of dexamethasone orally on days 1, 8, 15, and 22 (weekly). Ixazomib will be administered 4mg orally on days 1, 8 and 15.
  Interventions: Drug: Ixazomib; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Daratumumab-Hyaluronidase-Fihj@1,800 Mg-30,000 Unit/15 mL@SUBCUT@VIAL (ML)

INTERVENTIONS:
Drug: Ixazomib — 4mg PO days 1,8,15 on 28-day cycle
  Other Names: Ninlaro
Drug: Pomalidomide — 4mg days PO 1-21/28 days
  Other Names: Pomalyst
Drug: Dexamethasone — 40mg** PO weekly
  ** starting dose for age >75 may be 20mg
  Other Names: Decadron
Drug: Daratumumab-Hyaluronidase-Fihj@1,800 Mg-30,000 Unit/15 mL@SUBCUT@VIAL (ML) — 1800mg SQ weekly x 8 weeks, biweekly x 8 doses, then monthly
  Other Names: Darzalex Faspro

SUMMARY:
The purpose of this study is to determine the overall response rate of patients with Multiple Myeloma to the combination of Daratumumab, Ixazomib, Pomalidomide and Dexamethasone.

DETAILED DESCRIPTION:
The purpose of this study is to determine the overall response rate of patients with Multiple Myeloma to the combination of Daratumumab, Ixazomib, Pomalidomide and Dexamethasone.

The drugs being used in this study are daratumumab ixazomib, pomalidomide, and dexamethasone. Ixazomib may stop the growth of cancer by interfering with proteasomes (the protein breakdown mechanism in the cells). Pomalidomide, and dexamethasone are standard drugs that can change and regulate the immune system and may stop cancer cells from growing. Both Ixazomib and Daratumumab are approved for use in Multiple Myeloma, but not in this combination.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be registered into the mandatory POMALYST REMS program and be willing and able to comply with the requirements of the POMALYST REMS program.
* Confirmed diagnosis of Multiple Myeloma having received 1 and 3 prior lines of treatment
* Relapsed and/or refractory disease
* Measurable disease
* Life expectancy of more than 3 months
* ECOG performance status of 0, 1, or 2
* No prior progression on pomalidomide
* All pts must have received prior lenalidomide therapy and been determined to be relapsed and/or refractory.
* Adequate hepatic function
* Adequate renal function
* Additional Laboratory Requirements

  1. ANC ≥1.0 x 10^9/L, Hgb ≥8 g/dL (transfusion permitted)
  2. Platelet count ≥75 x 10^9/L (≥ 50x10^9/L if bone marrow plasma cells are ≥50% of cellularity)
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity from the time of signing the informed consent for through 120 days after the last dose of study medication.
* Women of childbearing potential have negative pregnancy test within 72 hours of initiating study drug dosing.
* Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential even if they have had a successful vasectomy starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the POMALYST REMS program.
* Subjects must agree to take enteric-coated aspirin 81 mg orally daily, or if history of prior thrombotic disease, must be fully anticoagulated with warfarin (INR 2-3) or be treated with full-dose, low molecular weight heparin, as if to treat deep venous thrombosis (DVT)/pulmonary embolism (PE) at the investigator's discretion.

Exclusion Criteria:

* Current or anticipated use of other investigational agents.
* Prior daratumumab or ixazomib use
* Patients who are refractory to pomalidom
* Non-secretory or hyposecretory multiple myeloma defined as:
* Plasma cell leukemia (>2.0 x 10 9/L circulating plasma cells by standard differential)
* Waldenström's macroglobulinemia or IgM myeloma
* Known central nervous system involvement by multiple myeloma
* Radiotherapy to multiple sites or immunotherapy within 2 weeks before enrollment (localized radiotherapy to a single site at least 1 week before start is permissible)
* Participation in an investigational therapeutic study within 3 weeks or within 5 drug half-lives (t1/2) prior to first dose, whichever time is greater. Non-interventional trials (i.e. observational trials) are permitted at any time point
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Major surgery within 3 weeks prior to first dose
* Myocardial infarction within 6 months prior to enrollment, NYHA (New York Heart Association) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
* Known or suspected HIV infection, known HIV seropositivity
* Active hepatitis infection
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Subjects with known or suspected light chain amyloidosis of any organ.
* Known allergies, hypersensitivity, or intolerance to monoclonal antibodies or human proteins, Daratumumab, or its excipients. or known sensitivity to mammalian-derived products.
* Has known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal
* Has known moderate or severe persistent asthma within the past 2 years per asthma guidelines
* Known gastrointestinal disease or procedure that could interfere with the oral absorption or tolerance of ixazomib or pomalidomide, including difficulty swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 2 years
  Anti-cancer response as defined by the International Uniform Response Criteria Consensus Recommendations
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 years
  Treatment-emergent Grade 2-5 adverse events (AEs) will be assessed using NCI CTCAE v4.03 toxicity criteria

SECONDARY OUTCOMES:
Clinical benefit rate | 2 years
  CBR: minimal response +ORR
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival (PFS) is defined as the duration of time from start of treatment until objective tumor progression or death
Time to progression | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Time to progression is defined as the duration of time from start of treatment until objective tumor progression.
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall survival is defined as the duration of time from start of treatment to death
Minimal Residual Disease (MRD) | 1 year
  Assessment on the presence of minimal residual disease for those in stringent complete response
Quality of life (QOL) scores | 2 years
  Cancer Therapy Satisfaction Questionnaire and EORTC QLQ-MY20

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Costello, MD, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - UCSD Moores Cancer Center, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No